CLINICAL TRIAL: NCT05203809
Title: Continuous Temperature Monitoring for tHe Early Recognition of Febrile Neutropenia in Haematological MALignancies (THERMAL)
Brief Title: Continuous Temperature Monitoring for tHe Early Recognition of Febrile Neutropenia in Haematological MALignancies
Acronym: THERMAL
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Malaghan Institute of Medical Research (Other)
Responsible Party: Sponsor
Other Study IDs: H21/161
Record Dates: First submitted 2021-11-22; First posted 2022-01-24 (Actual); Last update posted 2022-01-24 (Actual); Status verified 2022-01

CONDITIONS: Haematological Malignancy; Leukemia; Lymphoma; Myeloma; Temperature Change, Body
Keywords: temperature monitor; continuous; wireless; febrile neutropenia
MeSH Terms: conditions — Hematologic Neoplasms; Leukemia; Lymphoma; Neoplasms, Plasma Cell; Body Temperature Changes; Febrile Neutropenia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

GROUPS / COHORTS (1):
- Observation group: Group of participants wearing continuous temperature monitoring device
  Interventions: Device: TempTraq temperature monitor

INTERVENTIONS:
Device: TempTraq temperature monitor — All participants will wear both TempTraq temperature monitor and CORE temperature monitor.
  Other Names: CORE temperature monitor

SUMMARY:
The THERMAL study is a pilot study to determine feasibility of using two separate continuous skin temperature monitors during intensive treatment for haematological malignancies. It involves participants wearing both the TempTraq and CORE temperature devices for up to 14 days, and then assessing their feasibility and tolerability with quantitative, semiquantitative and qualitative methods.

DETAILED DESCRIPTION:
Patients with haematological malignancies such as leukaemia, lymphoma and myeloma often require intensive treatments such as chemotherapy, stem cell transplantation (either autologous or allogeneic) or CAR T-cell therapy. All these therapies can lead to a period of prolonged neutropenia, or low neutrophils, when they are at very high risk of serious bacterial infections. While other countries use routine prophylactic antibiotics, Australasian practice is to focus on prompt recognition and treatment of infections. There is clear evidence that early recognition and treatment of febrile neutropenia with antibiotics leads to improved outcomes, with each hour delay in antibiotic administration associated with an 18% increase in mortality.

Current practice is to detect fevers by both routine and symptom-based intermittent ear thermometer testing, with routine monitoring being approximately every four hours. However, neutropenic patients may not develop symptoms before manifesting a fever, meaning that continuous temperature monitoring could potentially lead to earlier recognition and treatment of febrile neutropenia.

This pilot study seeks to determine the feasibility of using two separate continuous skin temperature monitors during intensive treatment for haematological malignancies, in the inpatient and outpatient setting. If feasible, this could be used to increase the amount of treatments that can be safely performed as outpatients, as well as allowing earlier identification and treatment of febrile neutropenia.

The two proposed measuring devices are: 1. TempTraq adhesive temperature sensor, a skin temperature sensor which is applied to the axilla for 72 hours, then replaced; and 2. CORE temperature sensor, a rechargeable skin temperature sensor that is attached to the chest with a chest strap.

The TempTraq device is an FDA cleared class 2 medical device, while the CORE temperature monitor has received emergency FDA approval as a medical device in the context of the COVID-19 pandemic.

If these devices are demonstrated to be feasible, the technology could potentially be used to improve monitoring of immunosuppressed patients out of hospital, allowing patients to receive treatment out of hospital or closer to home. It may also allow earlier detection of febrile neutropenia, and reduce the mortality from this.

ELIGIBILITY:
Inclusion Criteria:

* Age 16-75 years
* Diagnosis of acute leukaemia, lymphoma or myeloma by consultant haematologist or multidisciplinary meeting discussion
* Undergoing treatment with either induction chemotherapy, autologous stem cell transplant, allogeneic stem cell transplant, or chimeric antigen receptor (CAR) T-cell therapy as part of their normal care.

Exclusion Criteria:

* Medical condition that would result in discomfort from the application of chest or axillary monitoring.
* Allergy to a component of the monitoring devices
* Diminished capacity or any circumstance that would prohibit them from understanding and providing informed consent in accordance with ICH-GCP (International Conference on Harmonisation, Good Clinical Practice) principles.

Ages: 16 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: This pilot study aims to recruit 15-20 participants undergoing treatment at Wellington Regional Hospital between November 2021 and June 2022. These will be patients with either acute leukaemia, lymphoma or myeloma that are requiring intensive treatment for their haematological malignancy, such as induction chemotherapy (e.g. doxorubicin/cytarabine for acute myeloid leukaemia), autologous stem cell transplantation, allogeneic stem cell transplantation or chimaeric antigen receptor (CAR) T-cell therapy. Their treatment may be delivered as an inpatient or outpatient (with outpatient treatment more likely in the setting of autologous stem cell transplantation or CAR T-cell therapy).
Sampling Method: Non-Probability Sample
Enrollment: 20 (Estimated)
Dates: Start 2021-11-18 (Actual); Primary Completion 2022-06-30 (Estimated); Study Completion 2022-06-30 (Estimated)

PRIMARY OUTCOMES:
Time device was worn | 14 days
  Percentage of time that both CORE and TempTraq were worn against total time available

SECONDARY OUTCOMES:
Device usability based on System Usability Scale questionnaire | 12 days
  Comparison of results from System Usability Scale (SUS) questionnaire for both devices at day 4, 8 and 12. The SUS is reported on a scale of 1-5, with 5 indicating the best response.
Participant interest in device, based on Intrinsic Motivation Index questionnaire | 12 days
  Comparison of results from Intrinsic Motivation Index questionnaires for both devices at day 4, 8 and 12. The IMI is reported on a 1-6 scale, with 6 in general indicating a better outcome (however several questions require the result to be reversed).
Participant preference for TempTraq or CORE device | 14 days
  Whether participant had a preference for once device over the other at completion of monitoring. This is to be indicated with a binary "TempTraq or CORE" question.
Comparability to intermittent ear thermometer data | 14 days
  Whether the TempTraq and CORE recordings correlated to intermittent ear thermometer recordings at the same timepoints (intermittent ear thermometers being the current standard of care).
Time between fever identification | 14 days
  Difference in time between fever identification via TempTraq and CORE temperature devices and intermittent ear thermometer
Rates of skin irritation or infection | 14 days
  Percentage of devices noted to have skin irritation or infection.
Participant age in years | 14 days
  Age in years, to be reported with median and range, to allow description of participant characteristics
Participant ethnicity | 14 days
  Participant self-identification of ethnicity, as per New Zealand Ministry of Health Ethnicity Data Protocols, Level 1 numbering hierarchy (as described in: https://www.health.govt.nz/publication/hiso-100012017-ethnicity-data-protocols)
Participant diagnosis | 14 days
  Histological classification of diagnosis, as per World Health Organisation classification of haematological malignancies.
Participant body mass index | 14 days
  Body mass index at enrolment in kg/m2, using height and weight.
Haematological treatment that participant is undergoing during study period | 14 days
  Haematological treatment, such as chemotherapy, cellular therapy e.g. CAR T-cell therapy, or stem cell therapy (whether allogeneic or autologous).

CONTACTS AND LOCATIONS:
Locations (1):
- Malaghan Institute of Medical Research, Wellington, New Zealand

REFERENCES:
- [Derived] Fyfe RC, Larsen M, Blud D, Weinkove R. Continuous temperature monitoring for the detection of fever in haemato-oncology patients: a pilot study of two wearable devices (THERMAL). Intern Med J. 2025 Nov;55(11):1928-1933. doi: 10.1111/imj.70199. Epub 2025 Sep 26. PMID 41001994